CLINICAL TRIAL: NCT01073475
Title: Global Network for Women's and Children's Health Research Maternal Newborn Health Registry
Brief Title: Maternal Newborn Health Registry
Acronym: MNH
Status: Recruiting | Type: Observational
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Responsible Party: Sponsor
Other Study IDs: CP MNH
Record Dates: First submitted 2010-02-21; First posted 2010-02-23 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy Outcome Trends in Low-resource Geographic Areas
Keywords: Pregnancy; Maternal mortality; Neonatal mortality; Stillbirth; Maternal Cause of Death; Neonatal Cause of Death
MeSH Terms: conditions — Maternal Death; Stillbirth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pregnant women: Pregnant women in the MNH cluster
  Interventions: Other: There is no intervention associated with the parent MNHR study. For the MNHR COVID sub-study, participants will be asked to provide a blood specimen at or near delivery.
- Male and Female Infants: Male and Female Infants delivered in the clusters
  Interventions: Other: There is no intervention associated with the parent MNHR study. For the MNHR COVID sub-study, participants will be asked to provide a blood specimen at or near delivery.

INTERVENTIONS:
Other: There is no intervention associated with the parent MNHR study. For the MNHR COVID sub-study, participants will be asked to provide a blood specimen at or near delivery. — There is no intervention associated with the parent MNHR study
  For the MNHR COVID sub-study, each woman will be asked to provide a blood specimen of approximately 3-5 cc at or near delivery (at delivery or 14 days after) to be tested for COVID-19 antibodies. The person collecting the specimen will be a trained member of the registry staff. The ZEUS ELISA SARS-CoV-2 IgG Test System will be used and run at each site. RTI International will provide central quality support of the analyses.

SUMMARY:
The primary purpose of this population-based study is to quantify and understand the trends in pregnancy outcomes in defined low-resource geographic areas over time, in order to provide population-based data on stillbirths, neonatal and maternal mortality.

DETAILED DESCRIPTION:
The purpose of the Global Network for Women's and Children's Health Research is to develop and test feasible, sustainable interventions to improve the outcome of women and children and to develop research capacity in resource-poor settings. Because most of the sites have weak health care systems, unacceptably high rates of maternal and neonatal mortality and lack birth and death registries, they lack precise data on outcomes and measures of care. Information from a vital registry system will allow the Global Network to document maternal and neonatal mortality, design trials to address the major causes of poor outcome, assess the outcome of our interventions, and ultimately disseminate the results as the basis of public health policy.

A sub-study to the Maternal Newborn Health Registry will be conducted to understand the prevalence of COVID-19 among pregnant women, the association between COVID-19 and pregnancy outcomes, and the Knowledge, Attitudes, and Practices of pregnant women related to COVID-19 and its prevention during pregnancy. Women who consent to participation in the MNHR COVID sub-study will provide a blood specimen at or near delivery to be tested for COVID-19 antibodies. Four Global Network sites (Guatemala, Bangladesh, Nagpur India and Pakistan) will also collect and analyze blood specimen from participants during antenatal care visits.

ELIGIBILITY:
Inclusion Criteria:

* Community-level

  * Appropriate for long-term registry data collection and the conduct of ongoing Global Network research
  * At least 300 deliveries per year
* Participant-level

  * Pregnant women intending to deliver within study cluster
  * Women who deliver within the study cluster
  * Women who reside in the community but are transferred for care at delivery

Exclusion Criteria:

* Participant-level

  * Opt out of consent to include data in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All pregnant women meeting participant-level criteria and the infant(s) from their pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 950000 (Estimated)
Dates: Start 2008-05 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Maternal mortality rate | 42 days post delivery
  Maternal mortality rate by site and cluster
Stillbirth rate | Delivery
  Stillbirth rate by site and cluster
Early neonatal mortality rate | 28 days post delivery
  ENM by site and by cluster

SECONDARY OUTCOMES:
Cause of maternal death at less than or equal to 42 days | 42 days post delivery
  Data collected by site and by cluster
Cause of neonatal death at less than or equal to 28 days | 28 days post delivery
  Data collected by site and by cluster
Prevalence of COVID-19 antibody positive results during pregnancy | At 12-14 week antenatal care visit, at delivery or 14 days after
  Data collected by site and by cluster
Fetal/neonatal outcomes (spontaneous abortion, stillbirth, birth weight (g), and fetal growth restriction, early (7-day) and late (28-day) neonatal death, cause of death, congenital infections, and malformations) associated with COVID-19 positivity | At delivery, 7 days post delivery and 28 days post delivery
  Data collected by site and by cluster
Maternal outcomes (rate of infection, timing of infection, types of symptoms, death, cause of death) associated with COVID-19 positivity | At delivery, 42 days post delivery
  Data collected by site and by cluster
Knowledge, attitudes, and practices of pregnant women related to COVID-19 infection during pregnancy | At the 12-14 week Antenatal Care visit
  Data collected by site and by cluster
Peri-partum and postpartum depression | At delivery and 6 weeks post-partum
  Data collected by site and by cluster

CONTACTS AND LOCATIONS:
Overall Officials: Marion Koso-Thomas, MD, Study Director — Center for Research for Mothers and Children (NICHD)
Locations (15):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Colorado Denver, Aurora, Colorado
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Boston University, Boston, Massachusetts
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Virgina, Charlottesville, Virginia
- ICDDRB, Dhaka, Bangladesh
- Kinshasa School of Public Health, Kinshasa, Democratic Republic of the Congo
- Institute for Nutrition of Central America and Panama (INCAP), Guatemala City, Departamento de Guatemala, Guatemala
- India (2):
  - Lata Medical Research Foundation, Nagpur, India
  - KLE Academy of Higher Education and Research, Belagavi, Karnataka
- The Aga Khan University, Karachi, Pakistan, Pakistan
- University Teaching Hospital, Lusaka, Zambia, Zambia

REFERENCES:
- [Derived] Austad KE, Rao SR, Hibberd PL, Patel AB. Trends and determinants of the use of episiotomy in a prospective population-based registry from central India. BMC Pregnancy Childbirth. 2024 Sep 12;24(1):598. doi: 10.1186/s12884-024-06762-y. PMID 39267006
- [Derived] Switchenko N, Shukla V, Mwenechanya M, Chomba E, Patel A, Hibberd PL, Ambalavanan N, Figueroa L, Mazariegos M, Krebs NF, Goudar SS, Derman R, Esamai F, Liechty EA, Bucher S, Saleem S, Goldenberg RL, Lokangaka A, Tshefu A, Bose CL, Koso-Thomas M, Tan S, Nolen T, McClure EM, Carlo WA. Neonatal Respiratory Support Utilization in Low- and Middle-Income Countries: A Registry-Based Observational Study. Neonatology. 2024;121(1):116-124. doi: 10.1159/000534777. Epub 2023 Dec 4. PMID 38048757
- [Derived] Figueroa L, Harrison M, Mazariegos M, Goudar S, Kavi A, Derman R, Patel A, Das P, Hibberd PL, Saleem S, Naqvi F, Goldenberg RL, Haque R, Billah SM, Petri WA Jr, McClure EM, Tan S, Krebs NF. Maternal and perinatal outcomes of women with vaginal birth after cesarean section compared to repeat cesarean birth in select South Asian and Latin American settings of the global network for women's and children's health research. Matern Health Neonatol Perinatol. 2023 Nov 1;9(1):13. doi: 10.1186/s40748-023-00169-x. PMID 37908009
- [Derived] Patel A, Bann CM, Thorsten VR, Rao SR, Lokangaka A, Tshefu Kitoto A, Bauserman M, Figueroa L, Krebs NF, Esamai F, Bucher S, Saleem S, Goldenberg RL, Chomba E, Carlo WA, Goudar S, Derman R, Koso-Thomas M, McClure E, Hibberd PL. Can the date of last menstrual period be trusted in the first trimester? Comparisons of gestational age measures from a prospective cohort study in six low-income to middle-income countries. BMJ Open. 2023 Sep 20;13(9):e067470. doi: 10.1136/bmjopen-2022-067470. PMID 37730415
- [Derived] Marete I, Ekhaguere O, Bann CM, Bucher SL, Nyongesa P, Patel AB, Hibberd PL, Saleem S, Goldenberg RL, Goudar SS, Derman RJ, Garces AL, Krebs NF, Chomba E, Carlo WA, Lokangaka A, Bauserman M, Koso-Thomas M, Moore JL, McClure EM, Esamai F. Regional trends in birth weight in low- and middle-income countries 2013-2018. Reprod Health. 2020 Dec 17;17(Suppl 3):176. doi: 10.1186/s12978-020-01026-2. PMID 33334365
- [Derived] Patel AB, Bann CM, Garces AL, Krebs NF, Lokangaka A, Tshefu A, Bose CL, Saleem S, Goldenberg RL, Goudar SS, Derman RJ, Chomba E, Carlo WA, Esamai F, Liechty EA, Koso-Thomas M, McClure EM, Hibberd PL. Development of the Global Network for Women's and Children's Health Research's socioeconomic status index for use in the network's sites in low and lower middle-income countries. Reprod Health. 2020 Dec 17;17(Suppl 3):193. doi: 10.1186/s12978-020-01034-2. PMID 33334359
- [Derived] Pusdekar YV, Patel AB, Kurhe KG, Bhargav SR, Thorsten V, Garces A, Goldenberg RL, Goudar SS, Saleem S, Esamai F, Chomba E, Bauserman M, Bose CL, Liechty EA, Krebs NF, Derman RJ, Carlo WA, Koso-Thomas M, Nolen TL, McClure EM, Hibberd PL. Rates and risk factors for preterm birth and low birthweight in the global network sites in six low- and low middle-income countries. Reprod Health. 2020 Dec 17;17(Suppl 3):187. doi: 10.1186/s12978-020-01029-z. PMID 33334356
- [Derived] Bauserman M, Thorsten VR, Nolen TL, Patterson J, Lokangaka A, Tshefu A, Patel AB, Hibberd PL, Garces AL, Figueroa L, Krebs NF, Esamai F, Nyongesa P, Liechty EA, Carlo WA, Chomba E, Goudar SS, Kavi A, Derman RJ, Saleem S, Jessani S, Billah SM, Koso-Thomas M, McClure EM, Goldenberg RL, Bose C. Maternal mortality in six low and lower-middle income countries from 2010 to 2018: risk factors and trends. Reprod Health. 2020 Dec 17;17(Suppl 3):173. doi: 10.1186/s12978-020-00990-z. PMID 33334343
- [Derived] Goudar SS, Goco N, Somannavar MS, Kavi A, Vernekar SS, Tshefu A, Chomba E, Garces AL, Saleem S, Naqvi F, Patel A, Esamai F, Bose CL, Carlo WA, Krebs NF, Hibberd PL, Liechty EA, Koso-Thomas M, Nolen TL, Moore J, Iyer P, McClure EM, Goldenberg RL, Derman RJ. Institutional deliveries and stillbirth and neonatal mortality in the Global Network's Maternal and Newborn Health Registry. Reprod Health. 2020 Dec 17;17(Suppl 3):179. doi: 10.1186/s12978-020-01001-x. PMID 33334337
- [Derived] Patel AB, Simmons EM, Rao SR, Moore J, Nolen TL, Goldenberg RL, Goudar SS, Somannavar MS, Esamai F, Nyongesa P, Garces AL, Chomba E, Mwenechanya M, Saleem S, Naqvi F, Bauserman M, Bucher S, Krebs NF, Derman RJ, Carlo WA, Koso-ThomasMcClure MEM, Hibberd PL. Evaluating the effect of care around labor and delivery practices on early neonatal mortality in the Global Network's Maternal and Newborn Health Registry. Reprod Health. 2020 Nov 30;17(Suppl 2):156. doi: 10.1186/s12978-020-01010-w. PMID 33256790
- [Derived] Bauserman M, Nowak K, Nolen TL, Patterson J, Lokangaka A, Tshefu A, Patel AB, Hibberd PL, Garces AL, Figueroa L, Krebs NF, Esamai F, Liechty EA, Carlo WA, Chomba E, Mwenechanya M, Goudar SS, Ramadurg U, Derman RJ, Saleem S, Jessani S, Koso-Thomas M, McClure EM, Goldenberg RL, Bose C. The relationship between birth intervals and adverse maternal and neonatal outcomes in six low and lower-middle income countries. Reprod Health. 2020 Nov 30;17(Suppl 2):157. doi: 10.1186/s12978-020-01008-4. PMID 33256784
- [Derived] McClure EM, Saleem S, Goudar SS, Garces A, Whitworth R, Esamai F, Patel AB, Tikmani SS, Mwenechanya M, Chomba E, Lokangaka A, Bose CL, Bucher S, Liechty EA, Krebs NF, Yogesh Kumar S, Derman RJ, Hibberd PL, Carlo WA, Moore JL, Nolen TL, Koso-Thomas M, Goldenberg RL. Stillbirth 2010-2018: a prospective, population-based, multi-country study from the Global Network. Reprod Health. 2020 Nov 30;17(Suppl 2):146. doi: 10.1186/s12978-020-00991-y. PMID 33256783
- [Derived] Saleem S, Naqvi F, McClure EM, Nowak KJ, Tikmani SS, Garces AL, Hibberd PL, Moore JL, Nolen TL, Goudar SS, Kumar Y, Esamai F, Marete I, Patel AB, Chomba E, Mwenechanya M, Bose CL, Liechty EA, Krebs NF, Derman RJ, Carlo WA, Tshefu A, Koso-Thomas M, Siddiqi S, Goldenberg RL. Neonatal deaths in infants born weighing >/= 2500 g in low and middle-income countries. Reprod Health. 2020 Nov 30;17(Suppl 2):158. doi: 10.1186/s12978-020-01013-7. PMID 33256782
- [Derived] Dhaded SM, Somannavar MS, Moore JL, McClure EM, Vernekar SS, Yogeshkumar S, Kavi A, Ramadurg UY, Nolen TL, Goldenberg RL, Derman RJ, Goudar SS. Neonatal deaths in rural Karnataka, India 2014-2018: a prospective population-based observational study in a low-resource setting. Reprod Health. 2020 Nov 30;17(Suppl 2):161. doi: 10.1186/s12978-020-01014-6. PMID 33256777
- [Derived] Figueroa L, Garces A, Hambidge KM, McClure EM, Moore J, Goldenberg R, Krebs NF. Prevalence of clinically-evident congenital anomalies in the Western highlands of Guatemala. Reprod Health. 2020 Nov 30;17(Suppl 2):153. doi: 10.1186/s12978-020-01007-5. PMID 33256772
- [Derived] McClure EM, Garces AL, Hibberd PL, Moore JL, Goudar SS, Saleem S, Esamai F, Patel A, Chomba E, Lokangaka A, Tshefu A, Haque R, Bose CL, Liechty EA, Krebs NF, Derman RJ, Carlo WA, Petri W, Koso-Thomas M, Goldenberg RL. The Global Network Maternal Newborn Health Registry: a multi-country, community-based registry of pregnancy outcomes. Reprod Health. 2020 Nov 30;17(Suppl 2):184. doi: 10.1186/s12978-020-01020-8. PMID 33256769
- [Derived] Patel A, Pusdekar YV, Prakash AA, Simmons E, Waikar M, Rao SR, Hibberd PL. Trends and determinants of increasing caesarean sections from 2010 to 2013 in a prospective population-based registry in eastern rural Maharashtra, India. BMJ Open. 2019 Aug 5;9(8):e024654. doi: 10.1136/bmjopen-2018-024654. PMID 31383691
- [Derived] Patel A, Prakash AA, Das PK, Gupta S, Pusdekar YV, Hibberd PL. Maternal anemia and underweight as determinants of pregnancy outcomes: cohort study in eastern rural Maharashtra, India. BMJ Open. 2018 Aug 8;8(8):e021623. doi: 10.1136/bmjopen-2018-021623. PMID 30093518
- [Derived] Saleem S, Tikmani SS, McClure EM, Moore JL, Azam SI, Dhaded SM, Goudar SS, Garces A, Figueroa L, Marete I, Tenge C, Esamai F, Patel AB, Ali SA, Naqvi F, Mwenchanya M, Chomba E, Carlo WA, Derman RJ, Hibberd PL, Bucher S, Liechty EA, Krebs N, Michael Hambidge K, Wallace DD, Koso-Thomas M, Miodovnik M, Goldenberg RL. Trends and determinants of stillbirth in developing countries: results from the Global Network's Population-Based Birth Registry. Reprod Health. 2018 Jun 22;15(Suppl 1):100. doi: 10.1186/s12978-018-0526-3. PMID 29945647
- [Derived] Dhaded SM, Somannavar MS, Jacob JP, McClure EM, Vernekar SS, Yogesh Kumar S, Kavi A, Ramadurg UY, Moore JL, Wallace DP, Derman RJ, Goldenberg RL, Goudar SS. Early pregnancy loss in Belagavi, Karnataka, India 2014-2017: a prospective population-based observational study in a low-resource setting. Reprod Health. 2018 Jun 22;15(Suppl 1):95. doi: 10.1186/s12978-018-0525-4. PMID 29945645
- [Derived] Patel A, Prakash AA, Pusdekar YV, Kulkarni H, Hibberd P. Detection and risk stratification of women at high risk of preterm birth in rural communities near Nagpur, India. BMC Pregnancy Childbirth. 2017 Sep 19;17(1):311. doi: 10.1186/s12884-017-1504-4. PMID 28927395
- [Derived] Patel AB, Prakash AA, Raynes-Greenow C, Pusdekar YV, Hibberd PL. Description of inter-institutional referrals after admission for labor and delivery: a prospective population based cohort study in rural Maharashtra, India. BMC Health Serv Res. 2017 May 19;17(1):360. doi: 10.1186/s12913-017-2302-4. PMID 28526027
- [Derived] Wang ME, Patel AB, Hansen NI, Arlington L, Prakash A, Hibberd PL. Risk factors for possible serious bacterial infection in a rural cohort of young infants in central India. BMC Public Health. 2016 Oct 19;16(1):1097. doi: 10.1186/s12889-016-3688-3. PMID 27760543
- [Derived] Hibberd PL, Hansen NI, Wang ME, Goudar SS, Pasha O, Esamai F, Chomba E, Garces A, Althabe F, Derman RJ, Goldenberg RL, Liechty EA, Carlo WA, Hambidge KM, Krebs NF, Buekens P, McClure EM, Koso-Thomas M, Patel AB. Trends in the incidence of possible severe bacterial infection and case fatality rates in rural communities in Sub-Saharan Africa, South Asia and Latin America, 2010-2013: a multicenter prospective cohort study. Reprod Health. 2016 May 24;13(1):65. doi: 10.1186/s12978-016-0177-1. PMID 27221099
- [Derived] Patel AB, Meleth S, Pasha O, Goudar SS, Esamai F, Garces AL, Chomba E, McClure EM, Wright LL, Koso-Thomas M, Moore JL, Saleem S, Liechty EA, Goldenberg RL, Derman RJ, Hambidge KM, Carlo WA, Hibberd PL. Impact of exposure to cooking fuels on stillbirths, perinatal, very early and late neonatal mortality - a multicenter prospective cohort study in rural communities in India, Pakistan, Kenya, Zambia and Guatemala. Matern Health Neonatol Perinatol. 2015 Jul 21;1:18. doi: 10.1186/s40748-015-0019-0. eCollection 2015. PMID 27057335
- [Derived] Bucher S, Marete I, Tenge C, Liechty EA, Esamai F, Patel A, Goudar SS, Kodkany B, Garces A, Chomba E, Althabe F, Barreuta M, Pasha O, Hibberd P, Derman RJ, Otieno K, Hambidge K, Krebs NF, Carlo WA, Chemweno C, Goldenberg RL, McClure EM, Moore JL, Wallace DD, Saleem S, Koso-Thomas M. A prospective observational description of frequency and timing of antenatal care attendance and coverage of selected interventions from sites in Argentina, Guatemala, India, Kenya, Pakistan and Zambia. Reprod Health. 2015;12 Suppl 2(Suppl 2):S12. doi: 10.1186/1742-4755-12-S2-S12. Epub 2015 Jun 8. PMID 26063483
- [Derived] Althabe F, Moore JL, Gibbons L, Berrueta M, Goudar SS, Chomba E, Derman RJ, Patel A, Saleem S, Pasha O, Esamai F, Garces A, Liechty EA, Hambidge K, Krebs NF, Hibberd PL, Goldenberg RL, Koso-Thomas M, Carlo WA, Cafferata ML, Buekens P, McClure EM. Adverse maternal and perinatal outcomes in adolescent pregnancies: The Global Network's Maternal Newborn Health Registry study. Reprod Health. 2015;12 Suppl 2(Suppl 2):S8. doi: 10.1186/1742-4755-12-S2-S8. Epub 2015 Jun 8. PMID 26063350
- [Derived] Pasha O, Goudar SS, Patel A, Garces A, Esamai F, Chomba E, Moore JL, Kodkany BS, Saleem S, Derman RJ, Liechty EA, Hibberd PL, Hambidge K, Krebs NF, Carlo WA, McClure EM, Koso-Thomas M, Goldenberg RL. Postpartum contraceptive use and unmet need for family planning in five low-income countries. Reprod Health. 2015;12 Suppl 2(Suppl 2):S11. doi: 10.1186/1742-4755-12-S2-S11. Epub 2015 Jun 8. PMID 26063346
- [Derived] McClure EM, Saleem S, Goudar SS, Moore JL, Garces A, Esamai F, Patel A, Chomba E, Althabe F, Pasha O, Kodkany BS, Bose CL, Berreuta M, Liechty EA, Hambidge K, Krebs NF, Derman RJ, Hibberd PL, Buekens P, Manasyan A, Carlo WA, Wallace DD, Koso-Thomas M, Goldenberg RL. Stillbirth rates in low-middle income countries 2010 - 2013: a population-based, multi-country study from the Global Network. Reprod Health. 2015;12 Suppl 2(Suppl 2):S7. doi: 10.1186/1742-4755-12-S2-S7. Epub 2015 Jun 8. PMID 26063292
- [Derived] Patel A, Bucher S, Pusdekar Y, Esamai F, Krebs NF, Goudar SS, Chomba E, Garces A, Pasha O, Saleem S, Kodkany BS, Liechty EA, Kodkany B, Derman RJ, Carlo WA, Hambidge K, Goldenberg RL, Althabe F, Berrueta M, Moore JL, McClure EM, Koso-Thomas M, Hibberd PL. Rates and determinants of early initiation of breastfeeding and exclusive breast feeding at 42 days postnatal in six low and middle-income countries: A prospective cohort study. Reprod Health. 2015;12 Suppl 2(Suppl 2):S10. doi: 10.1186/1742-4755-12-S2-S10. Epub 2015 Jun 8. PMID 26063291
- [Derived] Dhaded SM, Somannavar MS, Vernekar SS, Goudar SS, Mwenche M, Derman R, Moore JL, Patel A, Pasha O, Esamai F, Garces A, Althabe F, Chomba E, Liechty EA, Hambidge K, Krebs NF, Berrueta M, Ciganda A, Hibberd PL, Goldenberg RL, McClure EM, Koso-Thomas M, Manasyan A, Carlo WA. Neonatal mortality and coverage of essential newborn interventions 2010 - 2013: a prospective, population-based study from low-middle income countries. Reprod Health. 2015;12 Suppl 2(Suppl 2):S6. doi: 10.1186/1742-4755-12-S2-S6. Epub 2015 Jun 8. PMID 26063125
- [Derived] Bauserman M, Lokangaka A, Thorsten V, Tshefu A, Goudar SS, Esamai F, Garces A, Saleem S, Pasha O, Patel A, Manasyan A, Berrueta M, Kodkany B, Chomba E, Liechty EA, Hambidge K, Krebs NF, Derman RJ, Hibberd PL, Althabe F, Carlo WA, Koso-Thomas M, Goldenberg RL, Wallace DD, McClure EM, Bose CL. Risk factors for maternal death and trends in maternal mortality in low- and middle-income countries: a prospective longitudinal cohort analysis. Reprod Health. 2015;12 Suppl 2(Suppl 2):S5. doi: 10.1186/1742-4755-12-S2-S5. Epub 2015 Jun 8. PMID 26062992
- [Derived] Marete I, Tenge C, Chemweno C, Bucher S, Pasha O, Ramadurg UY, Mastiholi SC, Chiwila M, Patel A, Althabe F, Garces A, Moore JL, Liechty EA, Derman RJ, Hibberd PL, Hambidge K, Goldenberg RL, Carlo WA, Koso-Thomas M, McClure EM, Esamai F. Lost to follow-up among pregnant women in a multi-site community based maternal and newborn health registry: a prospective study. Reprod Health. 2015;12 Suppl 2(Suppl 2):S4. doi: 10.1186/1742-4755-12-S2-S4. Epub 2015 Jun 8. PMID 26062899
- [Derived] Goudar SS, Stolka KB, Koso-Thomas M, Honnungar NV, Mastiholi SC, Ramadurg UY, Dhaded SM, Pasha O, Patel A, Esamai F, Chomba E, Garces A, Althabe F, Carlo WA, Goldenberg RL, Hibberd PL, Liechty EA, Krebs NF, Hambidge MK, Moore JL, Wallace DD, Derman RJ, Bhalachandra KS, Bose CL. Data quality monitoring and performance metrics of a prospective, population-based observational study of maternal and newborn health in low resource settings. Reprod Health. 2015;12 Suppl 2(Suppl 2):S2. doi: 10.1186/1742-4755-12-S2-S2. Epub 2015 Jun 8. PMID 26062714
- [Derived] Pasha O, Saleem S, Ali S, Goudar SS, Garces A, Esamai F, Patel A, Chomba E, Althabe F, Moore JL, Harrison M, Berrueta MB, Hambidge K, Krebs NF, Hibberd PL, Carlo WA, Kodkany B, Derman RJ, Liechty EA, Koso-Thomas M, McClure EM, Goldenberg RL. Maternal and newborn outcomes in Pakistan compared to other low and middle income countries in the Global Network's Maternal Newborn Health Registry: an active, community-based, pregnancy surveillance mechanism. Reprod Health. 2015;12 Suppl 2(Suppl 2):S15. doi: 10.1186/1742-4755-12-S2-S15. Epub 2015 Jun 8. PMID 26062610
- [Derived] Page CM, Patel A, Hibberd PL. Does smoke from biomass fuel contribute to anemia in pregnant women in Nagpur, India? A cross-sectional study. PLoS One. 2015 May 29;10(5):e0127890. doi: 10.1371/journal.pone.0127890. eCollection 2015. PMID 26024473
- [Derived] Goudar SS, Carlo WA, McClure EM, Pasha O, Patel A, Esamai F, Chomba E, Garces A, Althabe F, Kodkany B, Sami N, Derman RJ, Hibberd PL, Liechty EA, Krebs NF, Hambidge KM, Buekens P, Moore J, Wallace D, Jobe AH, Koso-Thomas M, Wright LL, Goldenberg RL. The Maternal and Newborn Health Registry Study of the Global Network for Women's and Children's Health Research. Int J Gynaecol Obstet. 2012 Sep;118(3):190-3. doi: 10.1016/j.ijgo.2012.04.022. Epub 2012 Jun 26. PMID 22738806
- See also: The Global Network for Women's and Children's Health Research website contains information for the MNH Registry as well as other Global Network studies — http://gn.rti.org/

DOCUMENTS (2):
  • Study Protocol (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT01073475/Prot_001.pdf
  • Informed Consent Form (2016-11-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT01073475/ICF_000.pdf